CLINICAL TRIAL: NCT03215784
Title: Impact of Fish Oil or Probiotic Intake on Maternal Obesity and Molecular Biomarkers in the Placenta
Brief Title: Gestational Obesity and Interventions With Probiotics or Fish Oil Trial
Acronym: GOPROFIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Maternidade Escola da UFRJ (Unknown)
Responsible Party: Principal Investigator, Fátima Lúcia de Carvalho Sardinha, Professor, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LBqN
Record Dates: First submitted 2017-07-10; First posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Obesity; Pregnancy; Inflammation
Keywords: obesity; placenta; inflammation; fish oil; probiotics
MeSH Terms: conditions — Obesity; Inflammation | interventions — Fish Oils; Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Eutrophy Control (Placebo Comparator): Gelatin capsules a day, from 28ª week to 36ª week gestation.
  Interventions: Dietary Supplement: Placebo
- Eutrophy+ Probiotic (Experimental): Capsules gastro resistant containing 2.5 billions colony forming unit (UFC) Lactobacillus rhamnosus GG + 2.5 billions colony forming unit (UFC) Bifidobacterium bifidum a day, from 28ª week to 36ª week gestation
  Interventions: Dietary Supplement: Probiotic
- Obesity + Fish oil (Experimental): DHA (100 mg) + EPA (137 mg) a day, from 13ª week gestation to 36ª week gestation
  Interventions: Dietary Supplement: Fish Oil
- Obesity + Probiotic (Experimental): 2.5 billions colony forming unit (UFC) Lactobacillus rhamnosus GG + 2.5 billions colony forming unit (UFC) Bifidobacterium bifidum a day, from 28ª week to 36ª week gestation
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Fish Oil
  Arms: Obesity + Fish oil
Dietary Supplement: Probiotic
  Arms: Eutrophy+ Probiotic; Obesity + Probiotic
Dietary Supplement: Placebo
  Arms: Eutrophy Control

SUMMARY:
Obesity is one of the most concerning health issues in the modern world, especially due to its association with greater risk of developing a wide range of chronic diseases. Pre-gestational obesity may increase the chances of maternal and fetal morbimortality, such as gestational diabetes mellitus, preeclampsia, macrosomia and, even, fetal death. It may also lead to long term disorders, enhancing the risk of excessive adiposity and metabolic syndrome in later life and, thus, contributing to the maintenance of the obesity cycle and its health effects through the subsequent generations. Alterations in placental function are thought to be deeply involved in this scenario, however further research on its molecular and biological mechanisms is needed. During pregnancy, there is a physiological enhancement of the inflammatory state, marked by higher circulating cytokines and macrophage placental infiltration, which favors fetal nutrient supply and adequate growth; however, this response is exacerbated in women with pre-pregnancy obesity, leading to adverse outcomes. In this context, interventions aiming to reduce excessive inflammation may prevent or minimize the negative impact of pre-pregnancy obesity on both maternal and offspring's health. There is strong evidence suggesting an important role of n-3 LC-PUFA (EPA and DHA) on the attenuation and resolution of inflammatory states, besides influencing maternal lipid profile, fetal and infant adipogenesis and neurodevelopment. Additionally, the consumption of probiotic supplements during gestation seams to promote adequate maternal weight gain and improve the profile of inflammatory molecules secreted in the milk. Therefore, the nutritional interventions with fish oil, as a source of EPA and DHA, or probiotics, in women with pre-pregnancy obesity, may change the intrauterine environment and reduce the risk of both short and long term metabolic disorders. This study aims to investigate the metabolic and molecular changes promoted by gestational obesity and evaluate the effectiveness of different dietary interventions (fish oil or probiotic) on preventing or minimizing such alterations. We expect to contribute to the understanding of the physiological and molecular mechanisms underlying maternal obesity and its association with adverse pregnancy outcomes, associated with increased risk of chronic diseases in adulthood.

ELIGIBILITY:
Inclusion Criteria:

* aged between 19 and 40 years
* gestational age of 13 weeks;
* BMI prepregnancy greater than 29.9 and less than 40 kg / m² [ degrees obesity 1 and 2, according to the World Health Organization (WHO, 2002) ] or prepregnancy BMI between 18.5 and 24 9 kg / m² [ eutrophic ( WHO, 2002 ) ]
* be free of chronic diseases (hypertension , cardiovascular disease, type 2 diabetes , thyroid diseases , cirrhosis , chronic hepatitis and chronic renal failure
* be free of infectious and parasitic diseases
* present gestation single fetus
* not being a smoker
* do not consume alcoholic beverages
* do not consume supplement containing AG

Exclusion Criteria:

* receive confirmation of diagnosis of chronic noncommunicable diseases (except obesity) and / or infectious
* pregnant women who did not complete all the steps provided for in the study

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Association between maternal obesity and systemic Inflammation in the Mother and the Activation of Placental Inflammatory Pathways | 28 weeks
Association between fish oil intake in obese mothers and systemic Inflammation in the Mother and the Activation of Placental Inflammatory Pathways | 28 weeks
Investigation of the effects of fish oil supplementation on the metabolome of maternal serum, umbilical cord serum and placenta in obese pregnant women. | 28 weeks
  The metabolome of maternal serum, umbilical cord serum and placenta of obese and healthy pregnant women was analyzed by nuclear magnetic resonance.
Association between probiotic supplementation and bacterial colonization in the maternal intestinal and vaginal microbiota | 36 weeks
  Evaluation of the maternal intestinal and vaginal microbiota through the quantification of bacteria

SECONDARY OUTCOMES:
Association between maternal obesity and placental fatty acid transporter expression | 28 weeks
Association between fish oil intake in obese mothers and placental fatty acid transporter | 28 weeks
Association between maternal inflammatory status and pregnancy outcomes | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fátima Lúcia C Sardinha, PhD, Study Director — Instituto de Nutrição Josué de Castro/ UFRJ
Locations (1):
- Maternidade Escola da Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Reynolds RM, Allan KM, Raja EA, Bhattacharya S, McNeill G, Hannaford PC, Sarwar N, Lee AJ, Bhattacharya S, Norman JE. Maternal obesity during pregnancy and premature mortality from cardiovascular event in adult offspring: follow-up of 1 323 275 person years. BMJ. 2013 Aug 13;347:f4539. doi: 10.1136/bmj.f4539. PMID 23943697
- [Background] Lawlor DA, Relton C, Sattar N, Nelson SM. Maternal adiposity--a determinant of perinatal and offspring outcomes? Nat Rev Endocrinol. 2012 Nov;8(11):679-88. doi: 10.1038/nrendo.2012.176. Epub 2012 Sep 25. PMID 23007319
- [Background] Medanic D, Pucarin-Cvetkovic J. [Obesity--a public health problem and challenge]. Acta Med Croatica. 2012 Dec;66(5):347-55. Croatian. PMID 23814963
- [Background] Sirimi N, Goulis DG. Obesity in pregnancy. Hormones (Athens). 2010 Oct-Dec;9(4):299-306. doi: 10.14310/horm.2002.1280. PMID 21112860
- [Background] Ingelfinger JR, Nuyt AM. Impact of fetal programming, birth weight, and infant feeding on later hypertension. J Clin Hypertens (Greenwich). 2012 Jun;14(6):365-71. doi: 10.1111/j.1751-7176.2012.00660.x. Epub 2012 May 21. PMID 22672090
- [Background] Al-Gubory KH, Fowler PA, Garrel C. The roles of cellular reactive oxygen species, oxidative stress and antioxidants in pregnancy outcomes. Int J Biochem Cell Biol. 2010 Oct;42(10):1634-50. doi: 10.1016/j.biocel.2010.06.001. Epub 2010 Jun 19. PMID 20601089
- [Background] Jordan RG. Prenatal omega-3 fatty acids: review and recommendations. J Midwifery Womens Health. 2010 Nov-Dec;55(6):520-8. doi: 10.1016/j.jmwh.2010.02.018. PMID 20974414
- [Background] Teixeira TF, Collado MC, Ferreira CL, Bressan J, Peluzio Mdo C. Potential mechanisms for the emerging link between obesity and increased intestinal permeability. Nutr Res. 2012 Sep;32(9):637-47. doi: 10.1016/j.nutres.2012.07.003. Epub 2012 Sep 7. PMID 23084636
- [Background] Larque E, Gil-Sanchez A, Prieto-Sanchez MT, Koletzko B. Omega 3 fatty acids, gestation and pregnancy outcomes. Br J Nutr. 2012 Jun;107 Suppl 2:S77-84. doi: 10.1017/S0007114512001481. PMID 22591905
- [Background] Dugoua JJ, Machado M, Zhu X, Chen X, Koren G, Einarson TR. Probiotic safety in pregnancy: a systematic review and meta-analysis of randomized controlled trials of Lactobacillus, Bifidobacterium, and Saccharomyces spp. J Obstet Gynaecol Can. 2009 Jun;31(6):542-552. doi: 10.1016/S1701-2163(16)34218-9. PMID 19646321
- [Background] Rautava S, Collado MC, Salminen S, Isolauri E. Probiotics modulate host-microbe interaction in the placenta and fetal gut: a randomized, double-blind, placebo-controlled trial. Neonatology. 2012;102(3):178-84. doi: 10.1159/000339182. Epub 2012 Jul 6. PMID 22776980
- [Background] El-Bacha T, Midlej V, Pereira da Silva AP, Silva da Costa L, Benchimol M, Galina A, Da Poian AT. Mitochondrial and bioenergetic dysfunction in human hepatic cells infected with dengue 2 virus. Biochim Biophys Acta. 2007 Oct;1772(10):1158-66. doi: 10.1016/j.bbadis.2007.08.003. Epub 2007 Sep 15. PMID 17964123
- [Background] Chen B, Longtine MS, Sadovsky Y, Nelson DM. Hypoxia downregulates p53 but induces apoptosis and enhances expression of BAD in cultures of human syncytiotrophoblasts. Am J Physiol Cell Physiol. 2010 Nov;299(5):C968-76. doi: 10.1152/ajpcell.00154.2010. Epub 2010 Sep 1. PMID 20810912
- [Background] Challier JC, Basu S, Bintein T, Minium J, Hotmire K, Catalano PM, Hauguel-de Mouzon S. Obesity in pregnancy stimulates macrophage accumulation and inflammation in the placenta. Placenta. 2008 Mar;29(3):274-81. doi: 10.1016/j.placenta.2007.12.010. Epub 2008 Feb 11. PMID 18262644
- [Background] Gaccioli F, Lager S, Powell TL, Jansson T. Placental transport in response to altered maternal nutrition. J Dev Orig Health Dis. 2013 Apr;4(2):101-15. doi: 10.1017/S2040174412000529. PMID 25054676
- [Background] Frayling TM, Timpson NJ, Weedon MN, Zeggini E, Freathy RM, Lindgren CM, Perry JR, Elliott KS, Lango H, Rayner NW, Shields B, Harries LW, Barrett JC, Ellard S, Groves CJ, Knight B, Patch AM, Ness AR, Ebrahim S, Lawlor DA, Ring SM, Ben-Shlomo Y, Jarvelin MR, Sovio U, Bennett AJ, Melzer D, Ferrucci L, Loos RJ, Barroso I, Wareham NJ, Karpe F, Owen KR, Cardon LR, Walker M, Hitman GA, Palmer CN, Doney AS, Morris AD, Smith GD, Hattersley AT, McCarthy MI. A common variant in the FTO gene is associated with body mass index and predisposes to childhood and adult obesity. Science. 2007 May 11;316(5826):889-94. doi: 10.1126/science.1141634. Epub 2007 Apr 12. PMID 17434869
- [Background] Innis SM. Fatty acids and early human development. Early Hum Dev. 2007 Dec;83(12):761-6. doi: 10.1016/j.earlhumdev.2007.09.004. Epub 2007 Oct 24. PMID 17920214
- [Background] Burton GJ, Fowden AL. The placenta: a multifaceted, transient organ. Philos Trans R Soc Lond B Biol Sci. 2015 Mar 5;370(1663):20140066. doi: 10.1098/rstb.2014.0066. PMID 25602070
- [Background] Haghiac M, Basu S, Presley L, Serre D, Catalano PM, Hauguel-de Mouzon S. Patterns of adiponectin expression in term pregnancy: impact of obesity. J Clin Endocrinol Metab. 2014 Sep;99(9):3427-34. doi: 10.1210/jc.2013-4074. Epub 2014 May 5. PMID 24796925
- [Background] Aye IL, Lager S, Ramirez VI, Gaccioli F, Dudley DJ, Jansson T, Powell TL. Increasing maternal body mass index is associated with systemic inflammation in the mother and the activation of distinct placental inflammatory pathways. Biol Reprod. 2014 Jun;90(6):129. doi: 10.1095/biolreprod.113.116186. Epub 2014 Apr 23. PMID 24759787
- [Background] Mando C, Calabrese S, Mazzocco MI, Novielli C, Anelli GM, Antonazzo P, Cetin I. Sex specific adaptations in placental biometry of overweight and obese women. Placenta. 2016 Feb;38:1-7. doi: 10.1016/j.placenta.2015.12.008. Epub 2015 Dec 17. PMID 26907375
- [Background] Mezouar D, Merzouk H, Merzouk AS, Merzouk SA, Belarbi B, Narce M. In vitro effects of vitamins C and E, n-3 and n-6 PUFA and n-9 MUFA on placental cell function and redox status in type 1 diabetic pregnant women. Placenta. 2016 Jun;42:114-21. doi: 10.1016/j.placenta.2016.04.013. Epub 2016 Apr 15. PMID 27238721
- [Background] Wietrak E, Kaminski K, Leszczynska-Gorzelak B, Oleszczuk J. Effect of Docosahexaenoic Acid on Apoptosis and Proliferation in the Placenta: Preliminary Report. Biomed Res Int. 2015;2015:482875. doi: 10.1155/2015/482875. Epub 2015 Aug 3. PMID 26339616
- [Background] Luoto R, Laitinen K, Nermes M, Isolauri E. Impact of maternal probiotic-supplemented dietary counselling on pregnancy outcome and prenatal and postnatal growth: a double-blind, placebo-controlled study. Br J Nutr. 2010 Jun;103(12):1792-9. doi: 10.1017/S0007114509993898. Epub 2010 Feb 4. PMID 20128938
- [Background] Simpson MR, Dotterud CK, Storro O, Johnsen R, Oien T. Perinatal probiotic supplementation in the prevention of allergy related disease: 6 year follow up of a randomised controlled trial. BMC Dermatol. 2015 Aug 1;15:13. doi: 10.1186/s12895-015-0030-1. PMID 26232126
- [Background] Lindsay KL, Kennelly M, Culliton M, Smith T, Maguire OC, Shanahan F, Brennan L, McAuliffe FM. Probiotics in obese pregnancy do not reduce maternal fasting glucose: a double-blind, placebo-controlled, randomized trial (Probiotics in Pregnancy Study). Am J Clin Nutr. 2014 Jun;99(6):1432-9. doi: 10.3945/ajcn.113.079723. Epub 2014 Mar 19. PMID 24646819
- [Background] Lindsay KL, Walsh CA, Brennan L, McAuliffe FM. Probiotics in pregnancy and maternal outcomes: a systematic review. J Matern Fetal Neonatal Med. 2013 May;26(8):772-8. doi: 10.3109/14767058.2012.755166. Epub 2013 Jan 11. PMID 23205866
- [Background] Barrett HL, Dekker Nitert M, Conwell LS, Callaway LK. Probiotics for preventing gestational diabetes. Cochrane Database Syst Rev. 2014 Feb 27;2014(2):CD009951. doi: 10.1002/14651858.CD009951.pub2. PMID 24574258
- [Background] Vitali B, Cruciani F, Baldassarre ME, Capursi T, Spisni E, Valerii MC, Candela M, Turroni S, Brigidi P. Dietary supplementation with probiotics during late pregnancy: outcome on vaginal microbiota and cytokine secretion. BMC Microbiol. 2012 Oct 18;12:236. doi: 10.1186/1471-2180-12-236. PMID 23078375
- [Background] Cho I, Blaser MJ. The human microbiome: at the interface of health and disease. Nat Rev Genet. 2012 Mar 13;13(4):260-70. doi: 10.1038/nrg3182. PMID 22411464
- [Result] Pinto J, Barros AS, Domingues MR, Goodfellow BJ, Galhano E, Pita C, Almeida Mdo C, Carreira IM, Gil AM. Following healthy pregnancy by NMR metabolomics of plasma and correlation to urine. J Proteome Res. 2015 Feb 6;14(2):1263-74. doi: 10.1021/pr5011982. Epub 2015 Jan 6. PMID 25529102
- [Result] Lindsay KL, Hellmuth C, Uhl O, Buss C, Wadhwa PD, Koletzko B, Entringer S. Longitudinal Metabolomic Profiling of Amino Acids and Lipids across Healthy Pregnancy. PLoS One. 2015 Dec 30;10(12):e0145794. doi: 10.1371/journal.pone.0145794. eCollection 2015. PMID 26716698
- [Result] Chen R, Zhou L, Dong J, Miao LY. A rapid and underivatized method for the determination of glutamine in human serum with ultra performance liquid chromatography-tandem mass spectrometry and its application. Int J Food Sci Nutr. 2015 May;66(3):243-7. doi: 10.3109/09637486.2014.986074. Epub 2015 Jan 13. PMID 25582177
- [Result] Araujo JR, Correia-Branco A, Ramalho C, Goncalves P, Pinho MJ, Keating E, Martel F. L-methionine placental uptake: characterization and modulation in gestational diabetes mellitus. Reprod Sci. 2013 Dec;20(12):1492-507. doi: 10.1177/1933719113488442. Epub 2013 May 7. PMID 23653387
- [Result] Kurpad AV, Anand P, Dwarkanath P, Hsu JW, Thomas T, Devi S, Thomas A, Mhaskar R, Jahoor F. Whole body methionine kinetics, transmethylation, transulfuration and remethylation during pregnancy. Clin Nutr. 2014 Feb;33(1):122-9. doi: 10.1016/j.clnu.2012.12.016. Epub 2013 Jan 11. PMID 23356955
- [Result] Pusukuru R, Shenoi AS, Kyada PK, Ghodke B, Mehta V, Bhuta K, Bhatia A. Evaluation of Lipid Profile in Second and Third Trimester of Pregnancy. J Clin Diagn Res. 2016 Mar;10(3):QC12-6. doi: 10.7860/JCDR/2016/17598.7436. Epub 2016 Mar 1. PMID 27134947
- [Result] Tibbetts AS, Appling DR. Compartmentalization of Mammalian folate-mediated one-carbon metabolism. Annu Rev Nutr. 2010 Aug 21;30:57-81. doi: 10.1146/annurev.nutr.012809.104810. PMID 20645850
- [Result] Yan J, Jiang X, West AA, Perry CA, Malysheva OV, Brenna JT, Stabler SP, Allen RH, Gregory JF 3rd, Caudill MA. Pregnancy alters choline dynamics: results of a randomized trial using stable isotope methodology in pregnant and nonpregnant women. Am J Clin Nutr. 2013 Dec;98(6):1459-67. doi: 10.3945/ajcn.113.066092. Epub 2013 Oct 16. PMID 24132975